CLINICAL TRIAL: NCT01753661
Title: A Parent-Directed, Multimedia Early Intervention Tool to Improve Outcomes in Underserved Children Who Are Deaf or Hard-of-Hearing
Brief Title: Project ASPIRE Efficacy Pilot: Achieving Superior Parental Involvement for Rehabilitative Excellence
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12-0125
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Parental Language Behaviors
Keywords: Hearing loss; Language; Behavior change; Early Intervention; Home visiting
MeSH Terms: conditions — Hearing Loss; Language | interventions — House Calls

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Project ASPIRE Treatment Condition (Experimental): The Project ASPIRE Treatment condition will receive the Project ASPIRE intervention program which includes the linguistic feedback reports and the multimedia education sessions. This group will complete the same assessments as the control group.
  Interventions: Behavioral: Linguistic Feedback Report; Behavioral: Multimedia Education Sessions
- EI-As-Usual Condition (Active Comparator): As an ethical decision, eligible participants may roll over to the experimental group after satisfactory completion of this treatment.
  Interventions: Behavioral: EI-As-Usual

INTERVENTIONS:
Behavioral: Linguistic Feedback Report — Throughout the study, parents will complete 16 total LENA recordings. The feedback report will include information on the parent's previous LENA recording(s), including the Adult Word Count (AWC), Conversational Turns (CTC), and TV Time (TVT). Parents in the treatment group will receive feedback reports for the baseline and 10 weekly recordings. Feedback reports will not be offered for the follow-up recordings
  Arms: Project ASPIRE Treatment Condition
Behavioral: Multimedia Education Sessions — Treatment group parents will receive 10 weekly home visit sessions (e.g. the ASPIRE Program) with an interventionist during which time they will review multimedia education modules. The sessions include feedback report review, module discussion, video modeling, and goal setting activities. The education modules provide parents with information on supporting the development of listening and spoken language for children with hearing loss.
  Other Names: Home Visits
  Arms: Project ASPIRE Treatment Condition
Behavioral: EI-As-Usual — The EI-as-usual condition will parallel the treatment condition. Families in the EI-as-usual condition will continue to receive their usual therapy. They will not participate in Project ASPIRE home visits or receive feedback on their recordings. Families in this group will complete the same assessments as the families in the treatment group.
  Arms: EI-As-Usual Condition

SUMMARY:
The purpose of the proposed exploratory research protocol is to investigate the feasibility and efficacy of Project ASPIRE, a parent-directed intervention aiming to increase parental skills and enrich children's early language environments and ultimately improve child outcomes in children with hearing loss from low-income backgrounds.

DETAILED DESCRIPTION:
We will test the curriculum's efficacy in increasing parental knowledge and skills with a pilot study funded by a U.S. Department of Education Institute for Education Sciences Goal 2 grant. We hypothesize that parents who complete the ASPIRE curriculum with an Early Intervention therapist will demonstrate enhanced understanding of their child's listening and language needs. This deeper understanding will support behavior changes that improve the language-learning environment through increased parental engagement and linguistic input. Knowledge increase and changes to the language environment will be apparent in comparative pre- vs. post-intervention assessment scores. In addition, child outcomes will demonstrate improved listening and spoken language trajectories.

To encourage behavior change and help parents track their progress, the curriculum will be coupled with "linguistic feedback" gathered by the Language Environment Analysis (LENA) recorders and software. With linguistic feedback, EI therapists and parents will be able to track the family's progress through skill building and set goals for behavior change. This feedback and goal setting will allow parents to translate their knowledge into behavior changes that enrich their child's early language environment.

ELIGIBILITY:
Inclusion Criteria:

* Child is under 4.5 years old
* Child uses at least one amplification device (hearing aid, cochlear implant, BAHA)
* Child has adequate amplification (at least 30 db in one ear)
* Parent speaks conversational English
* Family's communication choice includes spoken language
* Family is considered low-SES according to income and education proxies

Exclusion Criteria:

* Child is younger than 6 months of age
* Parent does not speak conversational English
* Child is over 4.5 years of age
* Family is considered high-SES according to income and education proxies

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Parental Behavior Change - Language ENvironment Analysis (LENA): Quantitative Linguistic Change | 16 recordings total over a 6 month period: Baseline (3 Recordings), Weeks 1-10, Week 14, Week 18, Week 22
  The Language Environment Analysis (LENA) system records the home audio environment of children with a recorder and processes the recording information with specialized computer software. Processed recordings provide information for researchers on the following adult language-related behaviors: Adult Word Count (AWC), Conversational Turn Count (CTC), Television Time (TVT), and Background Noise.
Child Behavior Change - LENA: Quantitative | 16 recordings over a 6 month period: Baseline (3 Recordings, approximately 1 per week for 3 weeks), Weeks 1-10, Week 14, Week 18, Week 22
  The LENA system provides information about child language behaviors in addition to adult language behaviors, including data for Child Vocalization Count (CVC) and Conversational Turn Count (CTC).

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression Screen, short form (CESD-10) | Approximately 3 weeks pre-intervention
  Validated brief depression screen for the parent. Parents who score above the cut score will be assessed for suicidal ideation and self harm. Appropriate referrals will be made following assessment.
MacArthur Child Development Inventories (CDIs) | Approximately 3 weeks pre-intervention; 3 months post-intervention
  Parent self-report of child expressive vocabulary.
Scale of Parental Involvement and Self-Efficacy (SPISE) | Approximately 3 weeks pre-intervention; 1 week post-intervention; 3 months post-intervention
  Parent self-report that assesses of self-efficacy relating to involvement in children's development.
Early Intervention Parenting Self-Efficacy Scale (EIPSES) | Approximately 3 weeks pre-intervention; 1 week post-intervention; 3 months post-intervention
  Parent self-report measure of self-efficacy relating to early intervention programs.
ASPIRE Knowledge Questionnaire | Approximately 3 weeks pre-intervention; 1 week post-intervention; 4 months post-intervention
  Questionnaire developed for use in the trial that assesses parent's knowledge of child development and hearing loss
Demographics | Approximately 3 weeks pre-intervention program
  Questionnaire about family background; child development history; child hearing loss and hearing devices
Parent Stress Index (PSI) | Approximately 3 weeks pre-intervention
  A self-report measure that assesses level of parenting-related stress
Little Ears | Approximately 3 weeks pre-intervention; 3 months post-intervention
  Short questionnaire about child's level of listening and language development following cochlear implant or hearing aid activation.
Ages and Stages Questionnaire (ASQ) | Approximately 3 weeks pre-intervention program
  A questionnaire concerning the child's development.
Child Behavior Checklist (CBCL) | Approximately 3 weeks pre-intervention
  Parent report of potentially problematic child behaviors.
Rosetti | Approximately 3 weeks pre-intervention; 3 months post-intervention
  Questionnaire assessing child's current language development
Capute Scales | Approximately 3 weeks pre-intervention
  Validated scales of child development.
Theories of Intelligence (TOI) | Approximately 3 weeks pre-intervention; 1 week post-intervention; 3 months post-intervention
  6-item questionnaire that assesses entity and incremental theories of intelligence.
Parental Behavior Change - LENA and Video: Qualitative Changes | Baseline (2 Visits), Week 10, Week 22
  LENA transcription:MLU, type/token, syntactical complexity, gesture Video: gesture, "responsive parenting"

CONTACTS AND LOCATIONS:
Overall Officials: Dana L Suskind, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States